CLINICAL TRIAL: NCT02471586
Title: ILUMIEN III: OPTIMIZE PCI: OPtical Coherence Tomography (OCT) Compared to Intravascular Ultrasound (IVUS) and Angiography to Guide Coronary Stent Implantation: a Multicenter RandomIZEd Trial in Percutaneous Coronary Intervention (PCI)
Brief Title: OPTIMIZE PCI: Multicenter Randomized Trial of OCT Compared to IVUS and Angiography to Guide Coronary Stent Implantation
Acronym: ILUMIEN III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJM-CIP-10034
Record Dates: First submitted 2014-11-17; First posted 2015-06-15 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Intravascular Ultrasound; Optical Coherence Tomography; SJM-CIP-10034
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrasonography, Interventional; Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: For those subjects randomized to the IVUS or Angiography treatment arms, the operating investigator at the site was blinded to the final post-PCI OCT run for the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (3):
- Coronary PCI guided by IVUS (Active Comparator): Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with IVUS guidance according to local standard practice. IVUS imaging is required pre and post stent implantation.
  At the end of the procedure, a final IVUS imaging run must be performed.
  After the final IVUS run, a blinded OCT imaging run shall be performed to document final stent dimensions and results.
  Interventions: Procedure: Coronary PCI guided by IVUS
- Coronary PCI guided by OCT (Active Comparator): Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with OCT guidance according to the algorithm described in the protocol. OCT imaging is required pre and post stent implantation.
  At the end of the procedure, a final OCT imaging run must be performed.
  Interventions: Procedure: Coronary PCI guided by OCT
- Coronary PCI guided by Angiography (Active Comparator): Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with angiography guidance according to local standard practice.
  At the end of the procedure, a blinded OCT shall be performed to document final stent dimensions and results.
  Interventions: Procedure: Coronary PCI guided by Angiography

INTERVENTIONS:
Procedure: Coronary PCI guided by IVUS — Imaging type
  Other Names: Intravascular Ultrasound
  Arms: Coronary PCI guided by IVUS
Procedure: Coronary PCI guided by OCT — Imaging type
  Other Names: Optical Coherence Tomography
  Arms: Coronary PCI guided by OCT
Procedure: Coronary PCI guided by Angiography — Imaging type
  Arms: Coronary PCI guided by Angiography

SUMMARY:
The objective of this clinical investigation is to demonstrate the safety and efficacy of an OCT guided strategy for stent implantation

DETAILED DESCRIPTION:
This is a prospective, post-market, international, multi-center, randomized clinical investigation in which the participants will be randomized in 1:1:1 ratio to undergo PCI with either OCT, IVUS, or Angiography guidance. The clinical investigation will be conducted at approximately 35 sites in the United States and outside the United States; approximately 25% of subjects will be enrolled in the United States.

Patients in the IVUS and OCT groups patients will undergo baseline and post PCI imaging with their randomized modality. In addition, the Angiography group and IVUS groups will undergo a blinded post-PCI OCT run to allow comparison of OCT derived minimum stent area (MSA) in both groups.

After hospital discharge, all patients will have clinical follow-up at 30 days, and 1 year.

ELIGIBILITY:
General Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient with an indication for PCI including:

   * Angina (stable or unstable),
   * Silent ischemia (a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present),
   * NSTEMI, or
   * Recent STEMI (>24 hours from initial presentation and stable).
3. Patients will undergo cardiac catheterization and possible or definite PCI with intent to stent using any non-investigational metallic drug-eluting stent (DES)
4. Signed written informed consent

Angiographic inclusion criteria:

1. The target lesion must be located in a native coronary artery with visually estimated reference vessel diameter of ≥2.25 mm to ≤3.50 mm.
2. Lesion length <40mm

General Exclusion Criteria:

1. Estimated creatinine clearance <30 ml/min using Cockcroft-Gault equation, unless the patient is on dialysis
2. STEMI within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital.
3. PCI within 24 hours preceding the study procedure.
4. PCI of a lesion within the target vessel within 12 months prior to the study procedure
5. Planned use of bare metal stent (BMS)
6. Planned use of bioresorbable vascular scaffold (BVS)
7. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP, at time of procedure.
8. Mobitz II second degree or complete heart block
9. Malignant ventricular arrhythmias requiring treatment
10. Pulmonary edema defined as patient with shortness of breath, evidence of volume overload on physical exam, and crepitations on physical exam (>1/3 of lungs) or radiographic interstitial or alveolar pulmonary edema
11. Subject is intubated.
12. Known LVEF <30%.
13. Severe valvular disease (e.g. severe mitral regurgitation or severe aortic stenosis)
14. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
15. Presence of one or more co-morbidities which reduces life expectancy to less than 12 months or may interfere with protocol study processes.
16. Known allergy to protocol-required concomitant medications including aspirin; clopidogrel, prasugrel, and ticagrelor; heparin and bivalirudin; or iodinated contrast that cannot be adequately pre-medicated.
17. Patient is participating in any other investigational drug or device clinical trial that has not reached its primary endpoint.
18. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within one week before treatment).

Angiographic Exclusion Criteria:

1. The presence of any non-study lesion in the target vessel with angiographic diameter stenosis >50%, or any additional target vessel stenosis which requires PCI either during or within 12 months after the study procedure
2. Left main diameter stenosis ≥30% or left main PCI planned.
3. Study target lesion in a bypass graft
4. Ostial RCA study target lesion
5. Chronic total occlusion (TIMI flow 0/1) study target lesion
6. Bifurcation study lesion with a planned dual stent strategy
7. In-stent restenosis study target lesion
8. Any study lesion characteristic resulting in the expected inability to deliver the IVUS or OCT catheter to the lesion pre and post PCI (e.g. moderate or severe vessel calcification or tortuosity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Ali, MD, Principal Investigator — Columbia Presbyterian Medical Center (NY); Gregg W Stone, MD, Study Chair — Columbia Presbyterian Medical Center (NY)
Locations (29):
- United States (17):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Scottsdale Healthcare Shea, Scottsdale, Arizona
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Heart Institute of Colorado, Broomfield, Colorado
  - Orlando Health, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - New York Presbyterian Hospital/Columbia University, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Eastern Cardiology, Greenville, North Carolina
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - St. Charles Medical Center, Bend, Oregon
  - Austin Heart, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The University of Texas Health Science at San Antonio, San Antonio, Texas
- Onze-Lieve-Vrouwziekenhuis Campus Aalst, Aalst, East Flanders, Belgium
- Klinikum der Justus-Liebig-Universität, Giessen, Hesse, Germany
- Italy (2):
  - Ospedale Papa Giovanni XXIII, Bergamo, Lombardy
  - Centro Cardiologico Monzino, Milan, Lombardy
- Japan (5):
  - Kobe University Hospital, Chuo-ku, Hyōgo
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
- Erasmus MC - Thoraxcenter, Rotterdam, South Holland, Netherlands
- Hospital Universitario de la Princesa, Madrid, Spain
- Kings College Hospital, Brixton, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali ZA, Karimi Galougahi K, Maehara A, Shlofmitz RA, Fabbiocchi F, Guagliumi G, Alfonso F, Akasaka T, Matsumura M, Mintz GS, Ben-Yehuda O, Zhang Z, Rapoza RR, West NEJ, Stone GW. Outcomes of optical coherence tomography compared with intravascular ultrasound and with angiography to guide coronary stent implantation: one-year results from the ILUMIEN III: OPTIMIZE PCI trial. EuroIntervention. 2021 Jan 20;16(13):1085-1091. doi: 10.4244/EIJ-D-20-00498. PMID 32540793
- [Derived] Ali ZA, Maehara A, Genereux P, Shlofmitz RA, Fabbiocchi F, Nazif TM, Guagliumi G, Meraj PM, Alfonso F, Samady H, Akasaka T, Carlson EB, Leesar MA, Matsumura M, Ozan MO, Mintz GS, Ben-Yehuda O, Stone GW; ILUMIEN III: OPTIMIZE PCI Investigators. Optical coherence tomography compared with intravascular ultrasound and with angiography to guide coronary stent implantation (ILUMIEN III: OPTIMIZE PCI): a randomised controlled trial. Lancet. 2016 Nov 26;388(10060):2618-2628. doi: 10.1016/S0140-6736(16)31922-5. Epub 2016 Oct 30. PMID 27806900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,759 subjects were initially consented, however only 450 subjects were actually randomized and enrolled into the trial across 29 sites. The first randomized subject was enrolled on May 13, 2015, and the last randomized subject was enrolled on April 5, 2016. Each site was allowed to enroll a maximum of 65 subjects in the trial. The subjects were followed through 12-months and the last subject follow-up visit was completed on April 25, 2017.
Pre-assignment Details: Of the 1759 subjects consented, 1309 subjects were not randomized due to failed screening (n=1230), roll-in subjects (n=74), withdrawal of consent (n=1), withdrawal by the investigator (n=3) and software malfunction (n=1).
Groups:
- Coronary PCI Guided by OCT: Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with OCT guidance according to the algorithm described in the protocol. OCT imaging is required pre and post stent implantation.
  At the end of the procedure, a final OCT imaging run must be performed.
  Coronary PCI guided by OCT: Imaging type
- Coronary PCI Guided by IVUS: Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with IVUS guidance according to local standard practice. IVUS imaging is required pre and post stent implantation.
  At the end of the procedure, a final IVUS imaging run must be performed.
  After the final IVUS run, a blinded OCT imaging run shall be performed to document final stent dimensions and results.
  Coronary PCI guided by IVUS: Imaging type
- Coronary PCI Guided by Angiography: Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with angiography guidance according to local standard practice.
  At the end of the procedure, a blinded OCT shall be performed to document final stent dimensions and results.
  Coronary PCI guided by Angiography: Imaging type
Period: Overall Study
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Started | 158 | 146 | 146
Completed | 153 | 136 | 142
Not Completed | 5 | 10 | 4
Not completed — Lost to Follow-up | 3 | 8 | 4
Not completed — Death | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography | Total
Number analyzed (Participants) | 158 | 146 | 146 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.3) | 65.8 (9.5) | 65.4 (11.2) | 65.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 39 | 39 | 127
  Male | 109 | 107 | 107 | 323
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 2 | 1 | 6
  Belgium | 1 | 2 | 1 | 4
  United States | 89 | 81 | 85 | 255
  Japan | 16 | 15 | 13 | 44
  Italy | 32 | 31 | 32 | 95
  United Kingdom | 4 | 4 | 3 | 11
  Germany | 4 | 3 | 3 | 10
  Spain | 9 | 8 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint (Powered): Post-PCI Median Minimum Stent Area (MSA)
Description: Post-PCI MSA will be assessed by OCT in each randomized arm, measured at the independent OCT core laboratory blinded to imaging modality assignment. Hierarchal manner testing will be as follows:
  1. Non-inferiority: OCT vs. IVUS guided stenting
     Non-inferiority of OCT guided stenting to IVUS guided stenting will be analyzed for the mean difference between the post PCI MSA for the OCT and IVUS arms with non-inferiority margin of 1.0 mm^2.
  2. Superiority: OCT vs. Angiography guided stenting
     If the OCT guided stenting arm was found to be non-inferior to the IVUS guided stenting arm, the superiority of OCT to angiography will be tested for the mean difference between the post PCI MSA for the OCT and angiography arms.
  3. Superiority: OCT vs. IVUS guided stenting
  If the OCT guided stenting arm was found to be superior to the IVUS guided stenting arm, then the superiority of OCT to IVUS will be tested for the mean difference between the post PCI MSA for the OCT and IVUS arms.
Time Frame: Post-procedure within 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
mm^2 | 5.79 [4.54 to 7.34] | 5.89 [4.67 to 7.80] | 5.49 [4.39 to 6.59]

2. Primary Outcome: Primary Safety Endpoint (Non-powered): Number of Participants With Procedural MACE (Major Adverse Cardiac Event)
Description: Procedural MACE defined as procedural complications (angiographic dissection, perforation, thrombus, and acute closure) requiring active interventions (prolonged balloon inflations, additional stent implantations, pericardiocentesis, thrombus aspiration and other).
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Participants
  Intra-Procedural Complications Required Active Interventions | 4 | 1 | 1
  Prolonged Balloon Inflations | 0 | 0 | 0
  Additional Stent implantation | 4 | 1 | 1
  Pericardiocentesis | 0 | 0 | 0
  Thrombus Aspiration | 0 | 0 | 0
  Other Interventions | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Acute Procedural Success
Description: Acute procedural success are classified as:
  A) Optimal (%)
  The MSA of the proximal segment is ≥95% of the proximal reference lumen area and the MSA of the distal segment is ≥95% of the distal reference lumen area.
  B) Acceptable (%)
  The MSA of the proximal segment is ≥90% and <95% of the proximal reference lumen area and the MSA of the distal segment is ≥90% and <95% of the distal reference lumen area.
  C) Optimal and Acceptable (%)
  The MSA of the proximal segment is ≥90% and <95% of the proximal reference lumen area and the MSA of the distal segment is ≥90% and <95% of the distal reference lumen area.
  D) Unacceptable (%)
  The MSA of the proximal segment is <90% of the proximal lumen area, and/or the MSA of the distal segment is <90% of the distal reference lumen area.
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
Participants
  Optimal (≥95%): number analyzed (Participants) | 140 | 130 | 136
  Optimal (≥95%) | 36 | 32 | 23
  Acceptable (90 to 95%) | 22 | 16 | 5
  Unacceptable (<90%) | 82 | 82 | 108

4. Secondary Outcome: Rate of Post-PCI Stent Expansion (%)
Description: Post-PCI stent expansion is defined as the minimum stent area divided by the average of proximal and distal reference lumen areas x 100.
Time Frame: Up to 1 hour post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage of stent expansion
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
percentage of stent expansion | 87.6 (16.6) | 86.5 (15.9) | 82.9 (12.9)

5. Secondary Outcome: Rate of Mean Stent Expansion (%)
Description: Mean stent expansion is defined as the mean stent area (stent volume/analyzed stent length) divided by the average of proximal and distal reference lumen areas x 100.
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Median (Inter-Quartile Range); unit: percentage of mean stent expansion
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
percentage of mean stent expansion | 105.8 [97.8 to 119.8] | 106.3 [96.7 to 116.6] | 101.4 [91.9 to 110.2]

6. Secondary Outcome: Number of Participants With Plaque Protrusion and Thrombus
Description: Plaque protrusion and thrombus is defined as a mass attached to the luminal surface or floating within the lumen, meeting the following criteria:
  Protrusion is defined as any mass at least 0.2 mm beyond the luminal edge of a strut and will be further classified as Major and Minor.
  Major: Protrusion area/Stent area at site of tissue protrusion ≥10%
  Minor: Protrusion area/Stent area at site of tissue protrusion<10%
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
Participants
  Major | 27 | 27 | 25
  Minor | 67 | 73 | 70

7. Secondary Outcome: Number of Participants With Untreated Reference Segment Disease
Description: Untreated reference segment disease is defined as untreated Mean Lumen Area (MLA) ≤60% of the adjacent reference segment lumen area up to 10 mm from the proximal and distal stent edges.
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
Participants | 44 | 45 | 39

8. Secondary Outcome: Number of Participants With Edge Dissections
Description: Edge Dissections are classified as
  A) Major (%): ≥60 degrees of the circumference of the vessel at site of dissection and/or ≥3 mm in length
  B) Minor (%): any visible edge dissection <60 degrees of the circumference of the vessel and < 3 mm in length
  C) All (Major and Minor)
  Edge dissections will be further classified as:
  I. Intimal (limited to the intima layer, i.e. not extending beyond the internal elastic lamina)
  II. Medial (extending into the media layer)
  III. Adventitial (extending through the external elastic membrane
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
Participants
  Major | 19 | 35 | 26
  Minor | 20 | 18 | 35
  All (Major and Minor) | 39 | 53 | 61
  Intimal | 16 | 11 | 21
  Medial | 27 | 45 | 40
  Adventitial | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Stent Malapposition
Description: Frequency (%) of incompletely apposed stent struts (defined as stent struts clearly separated from the vessel wall (lumen border/plaque surface) without any tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm and not associated with any side branch).
  Malapposition will be further classified as:
  Major: if associated with unacceptable stent expansion
  Minor: if not associated with significant under-expansion
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
Participants
  Major | 15 | 28 | 44
  Minor | 43 | 24 | 39
  All (Major and Minor) | 58 | 52 | 83

10. Secondary Outcome: Number of Participants With Border Detection (OCT Arm Only)
Description: The visibility of the vessel external elastic lamina (EEL) border by OCT will be evaluated at both reference sites (proximal and distal) and the MSA before AND after intervention and then classified into 3 grades:
  A) Good: ≥75% (270°) of visible circumference
  B) Moderate: ≥50% (180°) - <75% (270°) of visible circumference
  C) Poor: <50% (180°) of visible circumference
Time Frame: Pre-PCI OCT Run procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Groups:
- Coronary PCI Guided by IVUS: Intervention =Coronary stenting with planned drug eluting stent (DES). Stenting will be performed with IVUS guidance according to local standard practice.IVUS imaging is required pre and post stent implantation.
  At the end of the procedure, a final IVUS imaging run must be performed. After the final IVUS run, a blinded OCT imaging run shall be performed to document final stent dimensions and results.
  Coronary PCI guided by IVUS:Imaging type
- Coronary PCI Guided by Angiography: Intervention = Coronary stenting with planned drug eluting stent (DES). Stenting will be performed with angiography guidance according to local standard practice.
  At the end of the procedure, a blinded OCT shall be performed to document final stent dimensions and results.
  Coronary PCI guided by Angiography:Imaging type
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 144 | 0 | 0
Participants
  Poor <180º of Visible EEL Circumference | 7 | 0 | 0
  Moderate >=1800, <2700 of Visible EEL Circumference | 28 | 0 | 0
  Good >=2700 of Visible EEL Circumference | 109 | 0 | 0

11. Secondary Outcome: Number of Participants With Altered Clinical Decision Making on the Basis of the Post-stent Imaging Run
Description: Clinical decision making will be assessed on the basis of the post-stent imaging run
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 150 | 140 | 0
Participants
  OCT/IVUS Result Acceptable (Yes) | 53 | 78 | 0
  OCT/IVUS Result Acceptable (No) | 97 | 62 | 0

12. Secondary Outcome: Median Intra-stent Lumen Area (Intra-stent Flow Area)
Description: Intra-stent Lumen Area (Intra-stent Flow Area) is defined as stent area minus any protrusion
Time Frame: Up to 1 hour post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
mm^2 | 5.54 [4.34 to 7.05] | 5.71 [4.59 to 7.58] | 5.42 [4.25 to 6.36]

13. Secondary Outcome: Median Effective Lumen Area (Total Flow Area)
Description: Effective lumen area (Total flow area) is defined as Intra-stent Lumen Area plus any area of malapposition between the stent and the vessel wall (lumen border/plaque border).
Time Frame: Up to 1 hour post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 140 | 135 | 140
mm^2 | 5.68 [4.59 to 7.30] | 5.87 [4.76 to 7.59] | 5.52 [4.42 to 6.63]

14. Secondary Outcome: IVUS Secondary Endpoints: Comparison of Number of Participants With Dissection IVUS vs. OCT Imaging (IVUS Arm Only)
Description: Dissection (Major, Minimal, All) will be compared between IVUS and OCT Imaging cohorts
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 135 | 140 | 0
Participants
  Major: number analyzed (Participants) | 134 | 137 | 0
  Major | 35 | 15 | 0
  Minor: number analyzed (Participants) | 134 | 137 | 0
  Minor | 18 | 7 | 0
  All (Major and Minor): number analyzed (Participants) | 134 | 137 | 0
  All (Major and Minor) | 53 | 22 | 0

15. Secondary Outcome: IVUS Secondary Endpoints: Comparison of Number of Participants With Malapposition IVUS vs. OCT Imaging (IVUS Arm Only)
Description: Malapposition (Major, Minimal, All) will be compared between IVUS and OCT Imaging cohorts
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 135 | 140 | 0
Participants
  Major | 28 | 20 | 0
  Minor | 24 | 7 | 0
  All (Major and Minor) | 52 | 27 | 0

16. Secondary Outcome: IVUS Secondary Endpoints: Comparison of Number of Participants With Plaque or Thrombus Protrusion IVUS vs. OCT Imaging (IVUS Arm Only)
Description: Protrusion (Major, Minimal, All) will be compared between IVUS and OCT Imaging cohorts
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 135 | 140 | 0
Participants
  Major | 27 | 10 | 0
  Minor | 73 | 17 | 0
  All (Major and Minor) | 100 | 27 | 0

17. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Median Minimal Lumen Diameter
Description: Angiographic Endpoints (QCA) will be assessed as Minimal lumen diameter
Time Frame: Baseline
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm | 0.99 [0.70 to 1.24] | 1.03 [0.73 to 1.26] | 0.95 [0.68 to 1.21]

18. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Median Minimal Lumen Diameter
Description: Angiographic Endpoints (QCA) will be assessed as Minimal lumen diameter
Time Frame: Final Post-PCI, up to 1 hour after PCI procedure
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm
  In-stent | 2.71 [2.40 to 3.05] | 2.78 [2.54 to 3.09] | 2.71 [2.44 to 2.96]
  In-segment | 2.30 [2.03 to 2.59] | 2.41 [2.12 to 2.74] | 2.37 [2.11 to 2.60]

19. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Median Diameter Stenosis
Description: Angiographic Endpoints (QCA) will be assessed as diameter stenosis
Time Frame: Baseline
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: percentage of Diameter Stenosis
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
percentage of Diameter Stenosis | 64.1 [55.8 to 73.1] | 63.7 [56.0 to 73.0] | 66.0 [57.8 to 74.9]

20. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Median Diameter Stenosis
Description: Angiographic Endpoints (QCA) will be assessed as diameter stenosis
Time Frame: Final Post-PCI, up to 1 hour after PCI procedure
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: percentage of Diameter Stenosis
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
percentage of Diameter Stenosis
  In-stent | 5.0 [2.2 to 10.6] | 5.1 [2.6 to 8.6] | 6.2 [2.5 to 9.9]
  In-segment | 14.7 [9.6 to 22.9] | 13.4 [9.0 to 20.3] | 13.0 [8.7 to 18.2]

21. Secondary Outcome: Non OCT Secondary Endpoints (Angiographic Endpoints (QCA)) - Median Acute Lumen Gain Post-intervention
Description: Angiographic Endpoints (QCA) will be assessed as Acute lumen gain post-intervention
Time Frame: Final Post-PCI, up to 1 hour after PCI procedure
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm
  In-stent | 1.76 [1.45 to 2.05] | 1.75 [1.52 to 2.10] | 1.75 [1.48 to 2.04]
  In-segment | 1.32 [1.02 to 1.65] | 1.38 [1.15 to 1.71] | 1.36 [1.16 to 1.69]

22. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Median Maximum Stent Size/Reference Vessel Diameter Ratio
Description: Angiographic Endpoints (QCA) will be assessed as Maximum stent size/reference vessel diameter ratio. Maximum stent size refers to the largest stent diameter used in a treated segment. If only one stent was used, it is that stent diameter. If more than one stent were used, it is the larger of the stent diameters.
Time Frame: Baseline
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm | 2.78 [2.42 to 3.12] | 2.87 [2.56 to 3.17] | 2.76 [2.50 to 3.15]

23. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Median Maximum Stent Size/Reference Vessel Diameter Ratio
Description: as for outcome 22
Time Frame: Final Post-PCI, up to 1 hour after PCI procedure
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm | 2.82 [2.47 to 3.13] | 2.84 [2.58 to 3.17] | 2.72 [2.45 to 3.04]

24. Secondary Outcome: Non OCT Secondary Endpoints - Angiographic Endpoints (QCA): Number of Participants With Angiographic Dissection ≥ NHLBI Type B
Description: Angiographic Endpoints (QCA) will be assessed as Angiographic dissection ≥ NHLBI type B
Time Frame: Final Post-PCI, up to 1 hour after PCI procedure
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Participants | 1 | 1 | 1

25. Secondary Outcome: Procedural Endpoints (Site Reported): Median Total Stent Length
Description: Median Total Stent Length will be measured in millimeters.
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm | 23.5 [15.0 to 32.0] | 24.0 [16.0 to 32.0] | 20.0 [16.0 to 30.0]

26. Secondary Outcome: Procedural Endpoints (Site Reported): Median Stents Per Lesion
Description: Median Stents per lesion will be measured in counts
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: Stents per lesion
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Stents per lesion | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]

27. Secondary Outcome: Procedural Endpoints (Site Reported) - Median Maximal Stent Size
Description: Median Maximal stent size will be measured in millimeters.
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
mm | 3.00 [2.75 to 3.50] | 3.00 [2.75 to 3.50] | 3.00 [2.75 to 3.50]

28. Secondary Outcome: Procedural Endpoints (Site Reported) - Median Post-dilatation Inflations
Description: Post dilatation inflations will be assessed in terms of use of balloon inflations
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: Number of inflations
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Number of inflations | 2 [1 to 3] | 2 [1 to 3] | 1 [1 to 2]

29. Secondary Outcome: Procedural Endpoints (Site Reported): Median Maximum Inflation Pressure (Atm.)
Description: Median Maximum inflation pressure will be measured in atm.
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Median (Inter-Quartile Range); unit: atm
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
atm | 18 [16 to 20] | 20 [16 to 20] | 18 [16 to 20]

30. Secondary Outcome: Procedural Endpoints (Site Reported): Number of Participants With Additional Interventions
Description: Participants will be analyzed for the use of additional inventions
  Additional interventions used on the basis of the post stent imaging run will be either use of Larger Balloon, Use of Higher Inflation Pressures, Use of Additional Inflations, Use of Additional Stent(s), Thrombus Aspiration, or Other Interventions
Time Frame: During procedure, an average of 1 hour
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 0
Participants
  Larger Diameter Balloon: number analyzed (Participants) | 82 | 60 | 0
  Larger Diameter Balloon | 51 | 28 | 0
  Higher Pressure Balloon: number analyzed (Participants) | 82 | 60 | 0
  Higher Pressure Balloon | 57 | 40 | 0
  Additional Stent: number analyzed (Participants) | 82 | 60 | 0
  Additional Stent | 11 | 12 | 0
  Other interventions: number analyzed (Participants) | 82 | 60 | 0
  Other interventions | 1 | 1 | 0

31. Secondary Outcome: Additional Procedural and Clinical Endpoints: Number of Participants With Angiography Defined Procedural Success Rate
Description: Angiography defined procedural success rate is defined as a final lesion angiographic diameter stenosis <30% (QCA) and TIMI III flow (QCA) without dissection ≥ NHLBI type C, perforation, prolonged chest pain or ST segment elevation or depression changes (>30 minutes), or procedural death.
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Participants | 135 | 130 | 131

32. Secondary Outcome: Additional Procedural and Clinical Endpoints - Number of Participants With Device Success Rate
Description: Device success rate (site reported):
  Successful OCT or IVUS imaging obtained pre and post PCI in the respective arms (does not include blinded OCT runs in the IVUS and Angiography arms)
Time Frame: During procedure, an average of 1 hour
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Participants | 149 | 139 | 0

33. Secondary Outcome: Additional Procedural and Clinical Endpoints - Number of Participants With Target Lesion Failure (TLF)
Description: Target Lesion Failure (TLF) at 1 year defined as cardiovascular death, target vessel myocardial infarction, or ischemia driven target-lesion revascularization.
  Target lesion is defined as the lesion designated for randomization to OCT vs. IVUS vs. Angiography.
Time Frame: 1 year
Population: Full Analysis Set (FAS) consists of all randomized subjects assigned to treatment per randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 158 | 146 | 146
Participants | 4 | 6 | 2

34. Secondary Outcome: Additional Procedural and Clinical Endpoints - Number of Participants With Peri-procedural Myocardial Infarction
Description: Number of Participants With Periprocedural Myocardial Infarction will be assessed at 1 year
Time Frame: 1 Year
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 156 | 146 | 146
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Description: All-Cause Mortality and Serious Adverse Events were monitored and analyzed. Non-serious adverse event information was not monitored for this study.
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by IVUS | Coronary PCI Guided by Angiography
All-Cause Mortality (participants affected / at risk) | 2/158 | 2/146 | 0/146
Serious Adverse Events (participants affected / at risk) | 37/158 | 25/146 | 26/146
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coronary PCI Guided by OCT (N=158) | Coronary PCI Guided by IVUS (N=146) | Coronary PCI Guided by Angiography (N=146)
Bleeding (Blood and lymphatic system disorders) | 2 | 0 | 0
Coronary restenosis (Cardiac disorders) | 0 | 0 | 1
Unstable angina (Cardiac disorders) | 2 | 1 | 1
Coronary perforation (Cardiac disorders) | 0 | 1 | 0
Sustained ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Chest pain (Cardiac disorders) | 6 | 4 | 7
Angina pectoris (Cardiac disorders) | 1 | 3 | 1
Myocardial ischemia (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Allergic drug reaction (Immune system disorders) | 0 | 1 | 0
Pneumonia caused by Gram-Negative Bacilli (Infections and infestations) | 0 | 1 | 0
Pneumonia caused by Haemophilus Influenzae (Infections and infestations) | 0 | 0 | 1
Acute viral hepatitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
In-stent restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Trauma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyponatremia (Investigations) | 0 | 1 | 0
Elevated troponin (Investigations) | 0 | 1 | 0
Arm pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seizure/convulsions/epilepsy (Nervous system disorders) | 1 | 0 | 0
Transient ischemic attack (TIA) (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1
Urinary tract infections (Renal and urinary disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
VASC vessel perforation (Vascular disorders) | 1 | 0 | 0
Vascular dissection (Vascular disorders) | 0 | 0 | 1
Vasc pseudoaneurysm (Vascular disorders) | 2 | 0 | 0
Arterial hypertension/hypertension (Vascular disorders) | 0 | 1 | 0
Left main dissection (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No